CLINICAL TRIAL: NCT00205842
Title: A Phase IIIb, Multicenter, Double-Blind, Placebo-Controlled, Parallel Study of Alvimopan for the Management of Opioid-Induced Postoperative Bowel Dysfunction/Postoperative Ileus
Brief Title: Study of Alvimopan for the Management of Opioid-induced Postoperative Bowel Dysfunction/Postoperative Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3753-001; 14CL314 (Other: Sponsor protocol number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Ileus
MeSH Terms: conditions — Ileus | interventions — alvimopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alvimopan

SUMMARY:
Patients undergoing major abdominal surgery are at highest risk for developing Postoperative Ileus (POI), occurring in nearly all cases. Signs and symptoms of POI may include abdominal distention and bloating, persistent abdominal pain; nausea and/or vomiting; variable reduction of bowel sounds; delayed passage of or inability to pass flatus or stool; and inability to tolerate a solid diet. This study will test the ability of alvimopan 12 mg given 30 to 90 minutes before the scheduled start of surgery to hasten the recovery of GI function in patients having partial small or large bowel resections.

DETAILED DESCRIPTION:
Postoperative ileus (POI) can be thought of as temporary slowing down or stopping of bowel function and a slowing down of movement of contents of the intestines. Patients undergoing major abdominal surgery are at highest risk for developing POI, occurring in nearly all cases. Signs and symptoms of POI may include abdominal distention and bloating, persistent abdominal pain; nausea and/or vomiting; variable reduction of bowel sounds; delayed passage of or inability to pass flatus or stool; and inability to tolerate a solid diet. This study will test the ability of alvimopan 12 mg given 30 to 90 minutes before the scheduled start of surgery to hasten the recovery of GI function in patients having partial small or large bowel resections.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for a partial small/large bowel resection with primary anastomosis; all procedures must be performed completely by open laparotomy.
* Subject is scheduled to receive primary postoperative pain management with intravenous (i.v.) patient-controlled analgesia (PCA) opioids.

Exclusion Criteria:

* Subject is scheduled for a total colectomy, colostomy, ileostomy, any laparoscopic or laparoscopically-assisted procedure, or subject has a history of gastrectomy, total colectomy, short bowel syndrome, or multiple previous abdominal surgeries performed by open laparotomy.
* Subject has complete bowel obstruction.
* Subject is currently taking opioid analgesics or has taken more than three doses of opioids (oral or parenteral) within the previous 7 days prior to the day of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660
Dates: Start 2004-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Time to recovery of GI function, which will be the time to Recovery of both upper GI function (tolerating solid food), and lower GI recovery (first bowel movement). Referred to as GI2.

SECONDARY OUTCOMES:
Time to discharge order written, time to actual discharge, time to tolerate solid food and time to first bowel movement

CONTACTS AND LOCATIONS:
Overall Officials: Adolor Corporation, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (1):
- 50 Sites, Exton, Pennsylvania, United States

REFERENCES:
- [Result] Ludwig K, Enker WE, Delaney CP, Wolff BG, Du W, Fort JG, Cherubini M, Cucinotta J, Techner L. Gastrointestinal tract recovery in patients undergoing bowel resection: results of a randomized trial of alvimopan and placebo with a standardized accelerated postoperative care pathway. Arch Surg. 2008 Nov;143(11):1098-105. doi: 10.1001/archsurg.143.11.1098. PMID 19015469
- [Derived] Ludwig K, Viscusi ER, Wolff BG, Delaney CP, Senagore A, Techner L. Alvimopan for the management of postoperative ileus after bowel resection: characterization of clinical benefit by pooled responder analysis. World J Surg. 2010 Sep;34(9):2185-90. doi: 10.1007/s00268-010-0635-9. PMID 20526599